CLINICAL TRIAL: NCT03362528
Title: Database and Calibration of a Non-invasive Glucose Monitoring Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RSP Systems A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RSP-10
Record Dates: First submitted 2017-11-20; First posted 2017-12-05 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short term collection of IMD data (Experimental): Subjects will collect spectral raman data on WM3.4NR four times a day for 30 days distributed over a time period of 60 days. Each timepoints are conducted in duplicate. Spectral data will be compared to standard BG measurements.
  Interventions: Device: WM3.4NR
- Long term collection of IMD data (Experimental): Subjects will collect spectral raman data on WM3.4NR four times a day for the initial 30 days, distributed over a time period of 60 days. Subjects will for the remaining 60 days of measurements, distributed over 120 days collect spectral data twice a day. Each timepoints are conducted in duplicate. Spectral data will be compared to standard BG measurements.
  Interventions: Device: WM3.4NR

INTERVENTIONS:
Device: WM3.4NR — Investigational Medical Device collecting spectral raman data from tissue.

SUMMARY:
This clinical study has been launched to collect spectral raman data paired with validated glucose reference values in private homes of subjects.

DETAILED DESCRIPTION:
Subjects will collect 2-4 daily optical raman readings paired with capillary Blood Glucose comparator in own home with maintaining usual routines. Subjects will either collect data for 30 days during a 60 days period or collect data for 90 days during 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 years of age or older
* Diabetic (all types) patients

Exclusion Criteria:

* Pregnant women
* Subjects not able to understand and read Danish
* In investigator's opinion, subject is not able to follow instructions as specified in the protocol
* Subjects not able to hold hand/arm steadily
* Extensive skin changes, tattoos or diseases on probe application site
* Rejection by prescreening optical measurements
* Known allergy to medical grade alcohol used to disinfect skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Generation and validation of predictive algorithms for determining blood glucose levels | 7 months
  Collected spectral raman data will found the development of predictive algorithms for glucose determination. Performance of predictive models will be evaluated using the consensus error grid

CONTACTS AND LOCATIONS:
Overall Officials: Jan Erik Henriksen, MD, Principal Investigator — Odense University Hospital, Dpt. of Endocrinology M
Locations (1):
- Department of Endocrinology M, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No